CLINICAL TRIAL: NCT02042144
Title: Correlate - Safety and Effectiveness of Regorafenib in Routine Clinical Practice Settings
Brief Title: Safety and Effectiveness of Regorafenib
Acronym: Correlate
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16821; SV1302 (Other: Company internal)
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Neoplasms
Keywords: Neoplasms, Colorectal
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Stivarga (Regorafenib, BAY73-4506)

INTERVENTIONS:
Drug: Stivarga (Regorafenib, BAY73-4506) — Patients diagnosed with mCRC who have been previously treated with, or are not considered candidates for, other locally approved standard treatment(s) and for whom the decision has been made per investigator's routine treatment practice to prescribe regorafenib

SUMMARY:
This study is a prospective observational cohort study. The study will be conducted in routine clinical practice settings. It is planned to enroll 1000 patients with metastatic Colorectal Cancer (mCRC) who have been previously treated with other approved treatments for metastatic disease and for whom a decision has been made by the physician to treat with regorafenib according to local health authority approved label. It is the aim of this observational cohort study to further characterize safety and effectiveness of regorafenib in routine clinical practice setting. Healthcare resource utilization in the routine provision of care is becoming increasingly important from a health economics and outcomes research perspective. Therefore, another aim of this observational cohort study is to capture healthcare resource associated with the management of treatment emergent adverse events in the real world setting. The primary objective of this study is to further characterize safety of regorafenib use in routine clinical practice settings. The secondary objective of this study is to assess the effectiveness of regorafenib in routine clinical practice settings as measured by Overall Survival (OS), Progression Free Survival (PFS) and Disease control rate (DCR). Health Related Quality of Life (HRQoL) Data will be collected in applicable countries.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mCRC who have been previously treated with, or are not considered candidates for, other locally approved standard treatment(s) and for whom the decision has been made per investigator's routine treatment practice to prescribe regorafenib.

Exclusion Criteria:

* Patients participating in an investigational program with interventions outside of routine clinical practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with mCRC who have been previously treated with, or are not considered candidates for, other locally approved standard treatment(s) and for whom the decision has been made per investigator's routine treatment practice to prescribe regorafenib.
Sampling Method: Probability Sample
Enrollment: 1034 (Actual)
Dates: Start 2014-04-08 (Actual); Primary Completion 2017-08-19 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Incidence of all treatment-emergent adverse events (TEAE) - Patients will be monitored for TEAE using the NCI-CTCAE Version 4.3 | Up to 42 months

SECONDARY OUTCOMES:
Overall Survival (OS), OS is defined as the time interval from the start of regorafenib therapy to death, due to any cause. | Up to 42 months
Progression free survival (PFS) is defined as the time interval measured from the day of start with regorafenib treatment to (radiological or clinical) progression or death, whichever comes first. | Up to 42 months
Disease control rate (DCR) - DCR is defined as percentage of patients, whose best response was not progressive disease (i.e. CR, PR or SD). Stable disease must be at least 6 weeks in duration. | Up to 42 months
Quality of Life - HRQoL using PRO questionnaire EQ-5D (8) in applicable countries | Up to 42 months
Healthcare resource utilization | Up to 42 months
  Hospitalization (Date, Length), Concomitant medication and procedures and any other anticancer therapies

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (13):
- Multiple Locations, Argentina
- Multiple Locations, Austria
- Multiple Locations, Czechia
- Multiple Locations, Denmark
- Multiple Locations, France
- Multiple Locations, Italy
- Multiple Locations, Luxembourg
- Multiple Locations, Mexico
- Multiple Locations, Netherlands
- Multiple Locations, Singapore
- Multiple Locations, Spain
- Multiple Locations, Switzerland
- Multiple Locations, Taiwan

REFERENCES:
- [Derived] Cervantes A, Tabernero J, Garcia-Carbonero R, Sastre J, Feliu J, Carmen Guillen-Ponce, Paredes BG, Carral A, Munoz J. Regorafenib in patients with metastatic colorectal cancer in Spain: from clinical trials to real-world evidence. Future Oncol. 2024;20(20):1401-1413. doi: 10.1080/14796694.2024.2340422. Epub 2024 Jun 11. PMID 38861286
- [Derived] Yeh KH, Yang TS, Hsu TC, Tzu-Liang Chen W, Chen HH, Teng HW, Lin BW, Kuan FC, Chiang FF, Duann CW, Li YS, Lin MT, Fiala-Buskies S, Ducreux M, Wang JY. Real-world evidence of the safety and effectiveness of regorafenib in Taiwanese patients with metastatic colorectal cancer: CORRELATE Taiwan. J Formos Med Assoc. 2021 Nov;120(11):2023-2031. doi: 10.1016/j.jfma.2020.12.015. Epub 2021 Jan 7. PMID 33422398
- [Derived] Ducreux M, Petersen LN, Ohler L, Bergamo F, Metges JP, de Groot JW, Wang JY, Garcia Paredes B, Dochy E, Fiala-Buskies S, Cervantes A, O'Connor JM, Falcone A; CORRELATE Investigators. Safety and effectiveness of regorafenib in patients with metastatic colorectal cancer in routine clinical practice in the prospective, observational CORRELATE study. Eur J Cancer. 2019 Dec;123:146-154. doi: 10.1016/j.ejca.2019.09.015. Epub 2019 Nov 4. PMID 31698328